CLINICAL TRIAL: NCT01210742
Title: The Efficacy of Hylan G-F 20 (Synvisc One) Injections in the Routine Management of Patients With Early Osteoarthritis of the Knee -a Randomised Controlled Trial (Pilot)
Brief Title: The Efficacy of Viscosupplementation for Early Knee Osteoarthritis
Acronym: EVOKE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/H0604/33
Record Dates: First submitted 2010-09-24; First posted 2010-09-28 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viscosupplementation with routine management (Experimental)
  Interventions: Device: Synvisc One
- Routine management (Active Comparator): Routine management for knee OA (NICE guidelines)
  Interventions: Other: Routine management

INTERVENTIONS:
Device: Synvisc One — Single intra-articular injection of a 6 mL of Hylan G-F 20 at baseline
  Arms: Viscosupplementation with routine management
Other: Routine management — Routine non-operative management for knee OA (NICE guidelines)
  Arms: Routine management

SUMMARY:
Treatment for early osteoarthritis (OA) of the knee is an increasing problem yet much of the research into OA, to date, concentrates on predisposition, genetic and cellular aspects and the treatment of late stage disease (arthroplasty). Clinicians reviewing patients with early OA have great difficulty in recommending an appropriate and efficacious intervention.

The first line of treatment for patients with early OA is exercise, self-management and weight loss. These tools are suggested to minimize the need for higher risk treatments such as non-steroidal antiinflammatory drugs (NSAIDs) and surgery. Viscosupplementation using intra-articular injections of hyaluronan (Synvisc One) is a relatively new treatment. To date, the ideal patient for viscosupplementation has yet to be defined. It is not known whether incorporation of viscosupplementation into the overall clinical management will have beneficial influence for patients with early OA of the knee.

This study will generate rigorous pilot data to assess the need and inform a larger randomized controlled trial (RCT) assessing the efficacy of viscosupplementation. The study will be a single blind randomised RCT. 60 patients with documented early OA will be randomised into one of two groups; Group V will undergo "one shot" viscosupplementation using Synvisc One in addition to routine physiotherapy management for knee OA. Group No V (control) will have no viscosupplementation but will undergo similar routine management including physiotherapy management for knee OA. Outcome measures will include walking pain (The Western Ontario and McMaster Universities Arthritis Index-WOMAC), the overall WOMAC score, Oxford Knee Score (OKS), American Knee Society score (AKS), complications, activity level and patient satisfaction. Health economics will also be evaluated. Measurements will be recorded pre-intervention and at six months following treatment.

The risks associated with viscosupplementation are minimal. Considering the limited resources currently available in health care, if the latter is shown to have higher effectiveness than physiotherapy alone, in addition to patient benefit, there will be important health economic implications.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* Radiographic evidence of OA in the tibiofemoral compartment (minute or definite osteophytes and a measurable joint space)
* Pain on walking (Visual Analogue Scale 0-10). Minimum of 4 and maximum of 9.
* Oxford knee score (OKS) of above 12 but below 36 (0-48, 48 no problem)
* Pain score of 1, 2 or 3 on Q1 (pain) of OKS.
* Suitable for viscosupplementation

Exclusion Criteria:

* OKS of below 12 and above 36 (0-48, 48 no problem)
* Pain score of 0 or 4 on Q1 (pain) of OKS.
* Grade 3 or 4 patellofemoral degeneration (Kellgren-Lawrence classification).
* Grade 3 or 4 tibiofemoral degeneration (Kellgren-Lawrence classification).
* A clinically apparent tense effusion of the target knee.
* Significant valgus/varus deformities.
* Ligamentous laxity or meniscal instability.
* Viscosupplementation history in any joint in the past 9 months.
* Previous surgery at the target knee in the past 6 months.
* Concomitant inflammatory disease (rheumatoid arthritis) or other condition that affects the joints.
* Use of prohibited medication/treatment for chronic pain.
* Pregnancy or new mothers who are breastfeeding.
* Systemic or intra-articular injection of corticosteroids in any joint within 3 months prior to screening.
* Obvious cartilage defects producing mechanical symptoms (i.e. locking).
* Listed for a knee replacement procedure for osteoarthritis of the knee.
* Have a history of failed conservative treatment (exercise therapy, physiotherapy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Walking pain | 6 months

SECONDARY OUTCOMES:
Patient satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David J Beard, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Biomedical Research Unit (BRU), Oxford, England, United Kingdom